Informed consent form - Development and Validation of a System for the Prediction of Challenging Behaviors of People with Autism Spectrum Disorder Based on a Smart Shirt a mixed-method design

Document date: 09/04/2022

A letter to the parents

Dear Parents,

The topic:

We would like to ask your permission to include your child in a research project

investigating the prediction of challenging behaviors in children with Autism.

The research:

The research is conducted by Professor Meir Lotan and Dr. Moti Zwilling and was

authorized by the Ariel University ethical committee.

What is going to actually happen:

Your child will wear the special smart shirt (which can measure heart rate, breathing,

activity) for a week when awake. When wearing the shirt, you will be asked to fill in a

follow-up chart describing clam and agitating moments. The shirt is easy and

comfortable to wear and will not be used if the child resists wearing it.

What will happen later:

We will analyze the data (from your child as well data collected from other participants)

with machine learning programs. These programs will be used to design an algorithm

which will be used as a base for an application intended to predict challenging behaviors

before they happen.

We ensure that:

Your participation is completely voluntary, and you can withdraw from this research at

any time, even if you previously gave your approval to participate.

The data will be saved in a password-protected computer and will be deleted at the end

of the research project.

No personal details regarding your child or any other participant will never be published

at any format.

For further details you can contact Professor Meir Lotan: by cellular: 0545944157 or

by E-mail: meirlo@ariel.ac.il

Thank you

Professor Meir Lotan

| We the parents of: | | | | |
|---|---|---|---|---|
| Total d | | TD. | | |
| The mother | | ID: | | |
| The father | | ID | | |
| Name of participat | ID | ID | | Birth date |
| Address: | | | | |
| We agree that: | | | | |
| A)will take part in this research project; | | | | |
| B) the details of the research project has been explained to me by | | | | |
| , | ; | | 1 | • |
| C) the research was approved by the Ariel Ethical committee; | | | | |
| , | | | will participate in the | |
| above-mentioned research project; | | | | |
| E) the data collected will be kept in confidentiality and will be deleted after | | | | |
| the termination of the project; | | | | |
| F) no private details regarding my daughter will ever be published at any | | | | |
| context or forum; | | | | |
| Father's signiture | Mother's Si | Mother's Signiture | | Date |
| 8 | | | | |
| Researcher's signiture | | | | |
| Name of researcher | Signiture | | Date | |